CLINICAL TRIAL: NCT00706706
Title: A Single-Arm, Open-Label, Multi-Center, Phase Iv, Safety And Efficacy Study Of Sunitinib Malate As First-Line Systemic Therapy In Chinese Patients With Metastatic Renal Cell Carcinoma (Post Approval Commitment Study)
Brief Title: Safety And Efficacy Study Of Sunitinib Malate As First-Line Systemic Therapy In Chinese Patients With Metastatic Renal Cell Carcinoma
Acronym: MRCC RCC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181132
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2012-12-20 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: sunitinib Phase IV metastatic renal cell carcinoma Chinese
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sunitinib (Experimental): single agent sunitinib, single arm
  Interventions: Drug: Sunitinib Malate (SU011248)

INTERVENTIONS:
Drug: Sunitinib Malate (SU011248) — Subjects will receive treatment with sunitinib in repeated 6-week cycles (4 weeks on, 2 weeks off), at a starting dose of 50 mg.

SUMMARY:
To investigate safety and efficacy of single agent sunitinib malate as first-line systemic therapy in Chinese patients with metastatic renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma with metastases with a component of clear (conventional) cell histology that is not amenable to surgery.
* Evidence of unidimensionally measurable disease
* Male or female, 18 years of age or older.
* ECOG performance status 0 or 1.
* Resolution of all acute toxic effects
* Adequate organ function.

Exclusion Criteria:

* Renal cell carcinoma without any clear (conventional) cell component.
* Prior systemic therapy for metastatic disease of any kind of RCC, such as Interferon or Interleukin, chemotherapy, hormonal, investigational or targeted therapies. Patients may have received prior adjuvant therapy with Interferon and/or Interleukin if recurrence occurred > 6 months after adjuvant therapy completion.
* Major surgery or radiation therapy <4 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
* NCI CTCAE grade 3 hemorrhage <4 weeks of starting the study treatment.
* Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, or in situ cervical cancer.
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of brain or leptomeningeal disease on screening CT or MRI scan.
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, and 6 months for pulmonary embolism.
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range with medication.
* Ongoing cardiac dysrhythmias, atrial fibrillation, or prolongation of the QTc interval to >450 msec for males or >470 msec for females.
* Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy).
* Ongoing treatment with therapeutic doses of Coumadin (low dose Coumadin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Current treatment on another clinical trial.
* Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- China (8):
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Wuhan, Hubei
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Chongqing
  - Pfizer Investigational Site, Shanghai
  - Pfizer Investigational Site, Tianjin
  - Pfizer Investigational Site, Xi'an

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181132&StudyName=Safety%20And%20Efficacy%20Study%20Of%20Sunitinib%20Malate%20As%20First-Line%20Systemic%20Therapy%20In%20Chinese%20Patients%20With%20Metastatic%20Renal%20Cell%20Carcinoma

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: Sunitinib 50 milligram (mg) capsule orally once daily for 4 weeks followed by 2 weeks off-treatment period in cycles of 6 weeks until disease progression, unacceptable sunitinib-associated toxicity or withdrawal.
Period: Overall Study
Arm/Group | Sunitinib
Started | 105
Completed | 0
Not Completed | 105
Not completed — Death | 53
Not completed — Lost to Follow-up | 7
Not completed — Study endpoint had reached | 45

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib: Sunitinib 50 mg capsule orally once daily for 4 weeks followed by 2 weeks off-treatment period in cycles of 6 weeks until disease progression, unacceptable sunitinib-associated toxicity or withdrawal.
Arm/Group | Sunitinib
Number analyzed (Participants) | 105
Age Continuous [Mean (Standard Deviation); unit: Years] | 54.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Time in weeks from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline, Day 28 of Cycles 1, 2, 3, 4 and even cycles thereafter until disease progression or every 2 months until death (up to 88 weeks)
Population: Safety population included those participants who had taken at least one dose of the study drug.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 105
Weeks | 61.7 [45.1 to 106.3]

2. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed response were those that persisted on repeat imaging study at least 4 weeks after initial documentation of response. CR was defined as disappearance of all lesions (target and/or non target). PR were those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions, with non target lesions not increased or absent.
Time Frame: as for outcome 1
Population: Per protocol (PP) population included those participants who had the disease under study, measurable disease and an adequate baseline disease assessment and had taken at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 103
Percentage of participants | 31.1 [22.3 to 40.9]

3. Secondary Outcome: Overall Survival (OS)
Description: Time in weeks from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 7. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: as for outcome 1
Population: Safety population included those participants who had taken at least one dose of the study drug.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Sunitinib
Number analyzed (Participants) | 105
Weeks | 133.4 [94.1 to NA] — Upper limit of confidence interval was not estimable due to the high number of participants censored for survival.

4. Secondary Outcome: One Year Survival Probability
Description: One year survival probability was defined as the probability of survival at one year after the first dose of study treatment.
Time Frame: Baseline, Day 28 of Cycles 1, 2, 3, 4 and even cycles thereafter, every 2 months until death (up to 1 year)
Population: Safety population included those participants who had taken at least one dose of the study drug.
Measure: Number (95% Confidence Interval); unit: Percent chance of survival
Arm/Group | Sunitinib
Number analyzed (Participants) | 105
Percent chance of survival | 72.0 [62.3 to 79.7]

ADVERSE EVENTS:
Time Frame: AEs/SAEs: From signing of informed consent form up to 28 days after last dose
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 13/105
Other Adverse Events (participants affected / at risk) | 102/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=105)
Right ventricular dysfunction (Cardiac disorders) | 1
Death (General disorders) | 1
Disease progression (General disorders) | 3
Pneumonia (Infections and infestations) | 2
Blood creatinine increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=105)
Anaemia (Blood and lymphatic system disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 29
Lymphopenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 24
Hypothyroidism (Endocrine disorders) | 26
Eyelid oedema (Eye disorders) | 24
Abdominal distension (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 51
Dry mouth (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 19
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6
Haemorrhoids (Gastrointestinal disorders) | 7
Mouth ulceration (Gastrointestinal disorders) | 30
Nausea (Gastrointestinal disorders) | 15
Stomatitis (Gastrointestinal disorders) | 18
Toothache (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 10
Chest pain (General disorders) | 8
Face oedema (General disorders) | 24
Fatigue (General disorders) | 54
Mucosal inflammation (General disorders) | 6
Oedema (General disorders) | 8
Oedema peripheral (General disorders) | 13
Pyrexia (General disorders) | 9
Alanine aminotransferase increased (Investigations) | 17
Aspartate aminotransferase increased (Investigations) | 16
Blood bilirubin increased (Investigations) | 10
Blood calcium decreased (Investigations) | 9
Blood creatinine increased (Investigations) | 19
Blood glucose increased (Investigations) | 6
Blood phosphorus decreased (Investigations) | 6
Blood thyroid stimulating hormone increased (Investigations) | 26
Blood urea increased (Investigations) | 9
Blood uric acid increased (Investigations) | 8
Haemoglobin decreased (Investigations) | 39
Lymphocyte count decreased (Investigations) | 8
Lymphocyte count increased (Investigations) | 9
Neutrophil count decreased (Investigations) | 41
Platelet count decreased (Investigations) | 54
Thyroxine increased (Investigations) | 6
Weight decreased (Investigations) | 23
White blood cell count decreased (Investigations) | 55
Decreased appetite (Metabolism and nutrition disorders) | 45
Back pain (Musculoskeletal and connective tissue disorders) | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 13
Dysgeusia (Nervous system disorders) | 29
Headache (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 6
Proteinuria (Renal and urinary disorders) | 8
Genital rash (Reproductive system and breast disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Dermatitis (Skin and subcutaneous tissue disorders) | 7
Hair colour changes (Skin and subcutaneous tissue disorders) | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 67
Rash (Skin and subcutaneous tissue disorders) | 28
Skin discolouration (Skin and subcutaneous tissue disorders) | 14
Swelling face (Skin and subcutaneous tissue disorders) | 6
Yellow skin (Skin and subcutaneous tissue disorders) | 15
Hypertension (Vascular disorders) | 39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.